CLINICAL TRIAL: NCT02668965
Title: The Effects of Intrauterine Infusion of Human Chorionic Gonadotropin at the Time of Embryo Transfer on IVF/ICSI Outcomes: Randomized, Double-blind Controlled Study
Brief Title: The Effects of Intrauterine Infusion of hCG at the Time of Embryo Transfer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Savinee Boonsuk, Miss, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: Si701/2015
Record Dates: First submitted 2016-01-27; First posted 2016-01-29 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Infertility
Keywords: Clinical pregnancy rate
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- control (No Intervention): intrauterine infusion with standard embryo culture media 10 microliters before embryo transfer
- intrauterine hCG (Experimental): intrauterine infusion with hCG (500 IU) 10 microliters before embryo transfer
  Interventions: Procedure: Intrauterine hCG (pregnyl)

INTERVENTIONS:
Procedure: Intrauterine hCG (pregnyl)
  Arms: intrauterine hCG

SUMMARY:
The purpose of this study is to determine whether intrauterine hCG can improve the implantation rate and clinical pregnancy rate after embryo transfer in IVF/ICSI cycle.

DETAILED DESCRIPTION:
Patients at infertility clinic, siriraj hospital who come to start IVF/ICSI treatment cycle or endometrial preparation for embryo transfer are consiferes as eligible subjects.

On the day of embryo transfer (both fresh and frozen-thaw cycle), the subjects will be randomized to 2 groups.

1. control group: embryo transfer after intrauterine infusion with standard embryo culture media 4-7 minutes
2. study group: embryo transfer after intrauterine infusion with hCG (Pregnyl) 4-7 minutes

The patients will come back for serum beta-hCG measurement 2 weeks later after embryo transfer and other 2 weeks later for transvaginal ultrasound if beta-hCG is positive.

ELIGIBILITY:
Inclusion Criteria:

1. infertile women aged 18-43 years
2. indicated or willing for IVF/ICSI treatment or endometrial preparation for embryo transfer

Exclusion Criteria:

1. Azoospermic male partner
2. Failure to retrieve oocyte after controlled ovarian hyperstimulation
3. No embryo retrieved for transfer
4. Endometrial preparation failure

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-03 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 2 weeks after positive serum beta-hCG
  Transvaginal ultrasound to confirm number of intrauterine gestational sac and fetal heart beats

SECONDARY OUTCOMES:
Chemical pregnancy rate | 2 weeks after embryo transfer
  positive serum beta-hCG more than 3
Implantation rate | 2 weeks after positive serum beta-hCG
  number of intrauterine gestational sac / number of embryo transferred

CONTACTS AND LOCATIONS:
Locations (1):
- Infertility unit, Siriraj Hospital, Bangkok, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes